CLINICAL TRIAL: NCT03350646
Title: Low Versus High Volume of Culture Medium During Embryo Transfer: a Randomized Clinical Trial.
Brief Title: Does the Volume of the Embryo Culture Medium During Embryo Transfer Affects the IVF Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Georgios Sigalos, Embryologist Bsc, Msc, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B-74/30-10-2014
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Clinical Pregnancy Rate
Keywords: embryo transfer; volume; culture medium; loading the catheter; clinical pregnancy rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low volume (20-25 μl) (Other): Low volume (20-25 μl)
  Interventions: Other: Volume of medium during embryo transfer
- High volume (40-45 μl) (Other): High volume (40-45 μl)
  Interventions: Other: Volume of medium during embryo transfer

INTERVENTIONS:
Other: Volume of medium during embryo transfer

SUMMARY:
The aim of this study was to evaluate if higher volume (40-45μl VS 20-25 μl) of media used for embryo transfer affects the clinical outcomes in fresh IVF cycles.Patients who fulfilled the inclusion criteria and agreed to participate in the study, were randomized, on the day of the embryo transfer, into group A: low volume (20-25 μL) and group B: high volume (40-45 μL)

DETAILED DESCRIPTION:
The volume of culture medium used for embryo transfer is a variable that has been speculated to affect the IVF outcome. It is known that ultra high volume (>100 μl) of medium during embryo transfer may result in embryo expulsion out of the uterus or ectopic pregnancy. Similarly, some authors advocate that ultra low volume of transferring medium (<10 μl) may negatively affect pregnancy and implantation rates.

However small differences in the volume of the culture medium may favor the outcome of the embryo transfer. The aim of this study was to evaluate if the use higher volume (40-45μl VS 20-25 μl) of media used for embryo transfer affects the clinical outcomes in fresh IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 45y.o.
2. BMI≤36 kg/m2,
3. Baseline FSH concentration <15 IU/l,
4. Ovarian stimulation with the same GnRH antagonist protocol
5. Normal uterine cavity with endometrium thickness >7mm and trilaminar morphology at the Time of transfer and semen
6. Parameters of >1 million /ml motile spermatozoa with >4% physiological morphology -

Exclusion Criteria:

1. PGD cycles
2. Frozen -thaw cycles
3. Natural cycles or patients following different ovarian stimulation protocol were excluded from the study

   -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 25 days after embryo transfer
  Number of clinical pregnancies expressed per 100 embryo transfer cycles

SECONDARY OUTCOMES:
Implantation rate | 25 days after embryo transfer
  The number of gestational sacs observed divided by the number of embryos transferred.
Ongoing pregnancy rate | 20 weeks
  Number of pregnancies till 20 weeks of gestation expressed per 100 embryo transfer cycles

REFERENCES:
- [Derived] Sigalos GAlpha, Michalopoulos Y, Kastoras AG, Triantafyllidou O, Vlahos NF. Low versus high volume of culture medium during embryo transfer: a randomized clinical trial. J Assist Reprod Genet. 2018 Apr;35(4):693-699. doi: 10.1007/s10815-017-1099-8. Epub 2017 Dec 12. PMID 29234954